CLINICAL TRIAL: NCT04276272
Title: Investigation of Changes in Tumour Choline Metabolism in Estrogen-receptor Positive / HER2 Negative Breast Cancer Patients Treated With CDK4/6 Inhibitors and Endocrine Therapy
Brief Title: D4 Choline Breast PET/CT
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); ECMC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18HH4880; 249165 (Other: IRAS)
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: HER2-negative Breast Cancer; ER Positive Breast Cancer; Metastatic Breast Cancer
Keywords: PET/CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Imaging scan — PET/CT scan
  Other Names: [18F]D4-FCH-PET/CT

SUMMARY:
The aim of this study is to evaluate the effect of CDK4/6 inhibitor treatment on the tumour choline metabolism as determined by [18F]D4-FCH PET/ computed tomography(CT) in breast cancer and to determine the suitability of [18F]D4-FCH-PET/CT as a non-invasive, early imaging biomarker for therapy response following CDK4/6 inhibitor treatment.

DETAILED DESCRIPTION:
A target of 16 evaluable participants will be recruited to this study. Participants will have[18F]D4-FCH PET/CT imaging on each of 2 visits Scan 1: Baseline scan to be conducted prior to initiating standard of care CDK4/6 inhibitor-based therapy drug therapy.

Scan2: Early post-treatment scan to be conducted at 4-6 weeks after initiating therapy.

Each participant will provide written consent to take part in the study before they undergo screening assessments to confirm eligibility. On the day of imaging the participants will have a blood sample taken for circulating tumour DNA prior to the scan.

A single dose of [18F]D4-FCH IV will be administered to the participant followed by dynamic/ whole body imaging.

Optional tumour biopsies at baseline and after 4-6 weeks of CDK4/6 inhibitor treatment will be obtained, or if there is a suitable archival pre-treatment biopsy that has been taken within 18 months, this can be retrieved for baseline analysis.

Clinical data for progression/ survival followed up for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with a histological diagnosis of locally advanced or metastatic estrogen-receptor positive, HER2 negative breast cancer
2. Written informed consent prior to admission in the study.
3. Target lesion diameter of ≥15mm that has not been previously irradiated and is located outside the liver
4. Female patients aged ≥ 18 years of age
5. For all patients: histologically confirmed locally advanced/ metastatic breast cancer with a previous biopsy confirming hormone receptor and HER2 status
6. ECOG performance status 0-2
7. Negative urine pregnancy test (within 2 hours prior to injection of imaging agent) in women of child bearing age and willingness to use contraception (barrier, abstinence, non-hormonal) for 3 weeks after injection of [18F]D4-FCH
8. Life expectancy > 3months
9. Adequate organ function as judged by investigator to include:

   * Hb≥ 10g/L
   * Creatinine clearance ≥45ml/min
10. Patients must have been appropriately staged (which may include contrast enhanced CT/ FDG-PET/ MRI) within 42 days of study entry and additional imaging according to local standard of care

Exclusion Criteria:

1. Pregnant or lactating women
2. Evidence of significant medical condition or laboratory finding which, in the opinion of the Investigator, makes it undesirable for the patient to participate in the trial
3. Participants with severe claustrophobia or who are unable to lie flat or fit into the scanner (≥350 lbs (160 Kg))
4. Prior use within 14 days of enrolment or concurrent therapy with any other investigational agent
5. Patients classified as radiation workers
6. Patient has previously received treatment with CDK 4/6 inhibitors

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 16 participants with HER2 negative/ER positive metastatic breast cancer who will be having CDK 4/6 inhibitor/endocrine therapy
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
The change in tumour uptake of [18F]D4-FCH (standardized uptake at 60 min, fractional retention) after approximately 4-6 weeks of CDK4/6 inhibitor-based therapy in patients with locally advanced or metastatic breast cancer | Through scan completion 4-6 weeks
  PET/CT

SECONDARY OUTCOMES:
Semi-quantitative assessment of the effect of CDK4/6 inhibitor-based therapy on [18F]D4-FCH tumour and normal tissue dynamics. Uptake of [18F]D4-FCH in normal tissues, and tumour target and non-target lesions combined (dynamic/whole body scans) | Through study completion, an average 2.5 years
  PET/CT
Correlation of [18F]D4-FCH uptake with tumour size or FDG-PET or appropriate standard clinical imaging | Through study completion, an average 2.5 years
  PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kenny, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust/ Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No